CLINICAL TRIAL: NCT06492317
Title: A Prospective, Single-center, Phase II Clinical Study of First-line Treatment for HER2 (Human Epidermal Growth Factor Receptor 2) Overexpressing Advanced Gastric Cancer With Disitamab Vedotin in Combination With Cadonilimab
Brief Title: RC48 Plus AK104 as First-line Treatment for HER2-overexpressing Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yongxu Jia, Chief Physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2021-K006-001
Record Dates: First submitted 2024-06-30; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: HER2-positive Gastric Cancer
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab vedotin plus cadonilimab (Experimental): Disitamab vedotin: 2.5mg/kg, D1, ivdrip, Q2W (every 2 weeks) ; Cadonilimab: 6mg/kg, D1, ivdrip, Q2W (every 2 weeks) ; until progressive disease (PD) or intolerable toxicity
  Interventions: Drug: Disitamab Vedotin; Drug: Cadonilimab

INTERVENTIONS:
Drug: Disitamab Vedotin — Disitamab Vedotin: 2.5mg/kg, d1, ivdrip, Q2W (every 2 weeks)
  Other Names: RC48
Drug: Cadonilimab — Cadonilimab: 6mg/kg, d1, ivdrip, Q2W (every 2 weeks)
  Other Names: AK104

SUMMARY:
A single-arm, single-center phase II trial study to assess the efficacy and safety of disitamab vedotin plus cadonilimab as first-line therapy for HER2-overexpressing advanced stomach carcinoma

DETAILED DESCRIPTION:
This study is a prospective, single-arm, single-center phase II trial. The purpose of the trial is evaluated Disitamab Vedotin (RC48) plus Cadonilimab (AK104) as first-line therapy for HER2-overexpressing advanced stomach carcinoma, and also check the adverse events (AEs) when participants are administered the combination treatment regimen. This study will include patients with HER2-overexpressing, locally advanced unresectable or metastatic gastric/gastroesophageal junction cancer who have not previously received systemic treatment including chemotherapy, targeted therapy, and immunotherapy. Enrolled patients will be treated with disitamab vedotin (2.5mg/kg, D1, ivdrip, Q2W) combined with cadonilimab (6mg/kg, D1, ivdrip, Q2W) until progressive disease (PD) or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age: more than 18 years, gender is not limited;
2. Confirmed locally advanced or distant metastasis gastric or gastroesophageal junction adenocarcinoma that is inoperable by pathological examination;
3. Confirmed HER2 2+or 3+ by immunohistochemistry (IHC);
4. At least 1 measurable lesion as determined by RECIST 1.1;
5. There is no prior systematic treatment, or the patient has received neoadjuvant/adjuvant chemotherapy, and the disease progresses or relapses more than 6 months after the treatment;
6. Eastern Cooperative Oncology Group (ECOG)performance status of 0-1;
7. Adequate organ function:

   1. Bone marrow function: Hemoglobin count (HGB)≥80g/L;
   2. Neutrophil count (NE)≥1.5×109/L;
   3. White blood cell count (WBC)≥3.5×109/L;
   4. Platelet count (PLT)≥100×109/L；
   5. Liver function: i. Serum total bilirubin (TBIL)≤1.5×ULN; ii. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP)≤3×ULN, patients with liver metastasis≤5×ULN;
   6. Kidney function: Blood creatinine (Cr) ≤1.5×ULN or Cockcroft Gault formula ≥ 60 mL/min;
   7. Cardiac function: New York Heart Association (NYHA) classification<Grade 3; Left ventricular ejection fraction≥50%;
8. At least 3 months life expectancy ;
9. The female of childbearing age must have taken reliable contraceptive measures or conducted a negative pregnancy test (serum or urine) within 7 days before enrollment, and are willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the test drug; the male must agree to use appropriate methods of contraception during the trial and 8 weeks after the last administration of the trial;
10. Willing to join the study and signed an informed consent form (ICF) with good compliance and cooperation in follow-up.

Exclusion Criteria:

1. Allergy to any trial drug and its excipients, or serious allergy history, or contraindication of the trial drugs;
2. Uncontrollable cardiovascular and cerebrovascular events , such as:

   1. NYHA grade 2 or above heart failure;
   2. Unstable angina pectoris;
   3. Myocardial infarction occurred within 12 months;
   4. Supraventricular or ventricular arrhythmia with clinical significance needs treatment or intervention;
   5. Cerebral hemorrhage and cerebral infarction (except for lacunar cerebral infarction without symptoms and without treatment);
   6. Serious cardiovascular and cerebrovascular events occurred within 12 months; Uncontrolled hypertension, i.e. systolic blood pressure>140 mmHg or diastolic blood pressure>90 mmHg after treatment;
   7. A history of arterial thrombosis or deep vein thrombosis within 6 months , or with evidence of bleeding tendency or medical history within 2 months, regardless of the severity;
   8. Stroke event or transient ischemic attack occurred within 12 months.
3. Received systematic treatment with Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use for ascites control) before the first administration within 2 weeks;
4. A history of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, acute lung disease, or systemic disease with poor control (including but not limited to diabetes, hypertension, etc.);
5. A history of active immune deficiency or autoimmune diseases, including HIV positive, or others acquired or congenital immune deficiency diseases, or organ transplantation;
6. Severe chronic or active infection requires systemic antibacterial, antifungal or antiviral treatment, including tuberculosis infection. A history of active tuberculosis infection ≥ 1 year should also be excluded, unless proved has been completed appropriate treatment;
7. Brain metastasis or leptomeningeal metastasis;
8. Clinically significant pleural effusion, pericardial effusion or ascites should be drained for many times within 2 weeks before the first administration of the drugs;
9. Another clinically detectable primary malignant tumor at the time of recruitment, or other malignant tumors in the past 5 years (except for fully treated skin basal cell carcinoma or cervical carcinoma in situ);
10. Any major surgery was performed ≤ 28 days before the drugs administration;
11. History of allogeneic stem cell transplantation or organ transplantation;
12. Be suffering gastrointestinal diseases: uodenal ulcer, ulcerative colitis, intestinal obstruction and others at present; or other conditions that may cause gastrointestinal bleeding or perforation judged by the researchers; or history of intestinal perforation or fistula, but has not recovered after surgical treatment;
13. Live vaccine are inoculated within 4 weeks (inclusive) before the first administration of the drugs, not including seasonal influenza vaccines but intranasal vaccine;
14. Other factors may lead to the forced termination of this trial according to the judgment of the investigator, such as other serious diseases (including psychological and mental diseases) requiring combined treatment, serious laboratory examination abnormalities, and family or social factors, which may affect the safety of the subject, or the collection of data and samples;
15. Participating in other therapeutic clinical studies or using research instruments within 4 weeks before the first administration;
16. Others conditions do not meet the inclusion according to the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-06 (Estimated); Primary Completion 2026-07-06 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects

SECONDARY OUTCOMES:
duration of response (DOR) | 12 months after the last subject participating in
  DOR (per RECIST 1.1) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
disease control rate (DCR) | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD) in total subjects
time to response (TTR) | 12 months after the last subject participating in
  TTR (per RECIST 1.1) is defined as the time from the starting date of study drug to the first time complete response (CR) or partial response (PR)
progression-free survival (PFS) | 12 months after the last subject participating in
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first
overall survival (OS) | 12 months after the last subject participating in
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China